CLINICAL TRIAL: NCT01241734
Title: Phase I/II Study of Lenalidomide in Combination With Rituximab, Ifosfamide, Etoposide, and Carboplatin (RICER)
Brief Title: Study of Lenalidomide in Combination With RICE With Lenalidomide Maintenance Post-Auto Transplant for DLBCL
Acronym: RICER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001132 - RV-DLBCL-PI-0463
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Revlimid (Lenalidomide) in Combination (Experimental): Study of Lenalidomide in Combination with Rituximab, Ifosphamide, Etoposide, and Carboplatin (RICE-R) as Salvage Therapy with Single Agent Lenalidomide as Maintenance Therapy Post-Autologous Stem Cell Transplantation
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — Stage I:
  Cohort 1: RICE + Lenalidomide 10mg days 1-7 Cohort 2: RICE + Lenalidomide 15mg days 1-7 Cohort 3: RICE + Lenalidomide 20mg days 1-7 Cohort 4: RICE + Lenalidomide 25mg days 1-7
  Stage II:
  RICE + Lenalidomide at the MTD days 1-7
  Stage III:
  Lenalidomide 25mg days 1-21 every 28 days
  Other Names: Lenalidomide

SUMMARY:
The standard of care therapy for DLBCL in the relapsed setting is RICE with the plan for the patient to proceed to transplant. This protocol will add Revlimid to the first 7 days of the RICE therapy and again after transplant as maintenance. To improve over all outcome and survival.

Hypothesis is that combining lenalidomide with standard of care (RICE) may increase overall response rate thus increasing the number of patients able to proceed with autologous stem cell transplant. This in turn may translate into improved overall survival and progression free survival.

DETAILED DESCRIPTION:
This is a 3-Stage, phase I/II, single-arm, open-label study. The first and second stage of the study will assess the safety and efficacy of lenalidomide, rituximab, Ifosfamide, etoposide, and carboplatin (RICER) for the treatment of DLBCL patients in first relapse. The third stage of the study will assess the safety and efficacy of post-autologous stem cell transplantation (ASCT) lenalidomide maintenance in patients with DLBCL.

In stage I of the study, escalating doses of lenalidomide (10, 15, 20, and 25 mg daily x 7 days on Days 1-7) along with RICE therapy will be given to cohorts of subjects in a standard 3+3 design (see section 5.4.2 for dose escalation schema) until the maximum tolerated dose (MTD) has been determined.

In stage II, all subjects will be given RICE plus the MTD of lenalidomide. The starting dose of lenalidomide in Stage II will be modified for reduced renal function as outlined in Section 5.4.2.

In both stage I and stage II, subjects who have stable disease or progression of disease after 2 cycles of RICER will be taken off study. Subjects who achieve > PR to 2 cycles of RICER will receive a third cycle followed by stem cell collection and ASCT.

Each cycle is 14 days. Delays in initiating a new cycle are allowed up to 14 days for Stages I and II. The planned number of cycles is 3.

After the second cycle, restaging with positron emission tomography (PET) and computerized tomography (CT) scans is performed. Patients with progressive disease are removed from the study, chemosensitive patients (CR/Cru and PR) proceed with third cycle of RICER. Stem cell collection will be completed within 10-14 days after third cycle of RICER. HDCMT-autoSCT will be performed after patient recovers from stem cell collection toxicities. High dose chemotherapy (HDCMT) followed by autologous stem cell transplant (autoSCT) involves administration of chemotherapy with BCNU, Etoposide, Ara-C, Melphalan (BEAM) followed by infusion of autologous stem cells. Involved-field radiation to the sites of bulky disease will be allowed prior to HDCMT-SCT.

Stage III, after recovery from aSCT, but not to exceed 90 days all eligible subjects will receive lenalidomide maintenance therapy (po daily on Days 1-21 q28 days) for up to 1 year. Delays in initiating a new cycle up to 28 days are allowed in Stage III. Subjects will be followed for progression- free survival and overall survival for up to 2 years. The starting dose of lenalidomide maintenance treatment will be based on calculated creatinine clearance within 28 days prior to the start of lenalidomide maintenance

ELIGIBILITY:
Inclusion Criteria:Understand and voluntarily sign an informed consent form.

1. Age 18 years at the time of signing the informed consent form.
2. Able to adhere to the study visit schedule and other protocol requirements.
3. Histologically confirmed diffuse large B cell lymphoma
4. Relapsed or refractory after one prior therapeutic treatment for DLBCL. Refractory is defined as patients received adequate prior treatment and did not respond during treatment or progressed within 90 days of last treatment.
5. Measurable disease with at least on bidimensional lymph node or tumor mass >1.5 cm in the longest diameter that can be followed for response as a target lesion as measured by PET or CT
6. Histologically confirmed involvement of the bone marrow by DLBCL on the bone marrow biopsy without other measurable disease
7. Eligible for autologous stem cell transplant
8. All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least two weeks prior to treatment in this study.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 2 at study entry (see Appendix B).
10. Laboratory test results within these ranges:

    * Absolute neutrophil count >1000 /mm³
    * Platelet count > 50,000/mm³ (unless bone marrow is heavily infiltrated with underlying disease (50% or more) Calculated creatinine clearance of ≥ 60 mL/min by Cockroft-Gault formula (Appendix E) for patients enrolled into the phase I portion of the study (Stage I). Calculated creatinine clearance of ≥ 30 mL/min by Cockroft-Gault formula for patients enrolled into the phase II portion of the study (Stage II). See Section 5.4.2 for lenalidomide dose adjustment for calculated creatinine clearance > 30ml/min and < 60ml/min.
    * Total bilirubin < 1.5 x Upper Limit of Normal (ULN).
    * Aspartate Aminotransferase (SGOT) and Alanine Aminotransferase (SGPT) < 3 x ULN.
11. Disease free of prior malignancies for > 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
12. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
13. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International unit (mIU)/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix A: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
14. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid (ASA) may use warfarin or low molecular weight heparin).

    -

Exclusion Criteria: Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.

1. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
3. Evidence of laboratory tumor lysis syndrome (TLS) by Cairo-Bishop Definition of Tumor Lysis Syndrome. Subjects may be enrolled upon correction of electrolyte abnormalities.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Concurrent use of other nonprotocol anti-cancer agents or treatments.
8. Known positive for HIV or active infectious hepatitis, type B or C.
9. Refusal of autologous stem cell transplant.
10. Patients with active central nervous system involvement based on clinical evaluation. Previously treated central nervous system (CNS) involvement that has remained asymptomatic for more than ninety days is allowed if no active CNS disease present as confirmed by MRI or/and lumbar puncture.
11. Concurrent uncontrolled serious medical ort psychiatric conditions likely to interfere with participation in this clinical study, as judged by investigator.
12. Prior Lenalidomide exposure for more than 28 days.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana Feldman, MD, Principal Investigator — Hackensack Meridian Health
Locations (2):
- United States (2):
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2010-2015
Groups:
- Stage I, Cohort 1: RICE + Lenalidomide 10mg days 1-7
- Stage I, Cohort 2: RICE + Lenalidomide 15mg days 1-7
- Stage I, Cohort 3: RICE + Lenalidomide 20mg days 1-7
- Stage I, Cohort 4: RICE + Lenalidomide 25mg days 1-7
- Stage II: RICE + Lenalidomide 25mg (MTD) days 1-7
Period: Overall Study
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Started | 3 | 4 | 3 | 3 | 5
Completed | 1 | 2 | 2 | 1 | 2
Not Completed | 2 | 2 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 5 | 18
Age, Continuous [Median (Full Range); unit: years] | 70 [66 to 75] | 60 [52 to 62] | 64 [53 to 72] | 63 [46 to 65] | 51 [22 to 68] | 61.5 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A portion of the Stage II patients were enrolled at an external site and some demographic details of these patients are no longer available.
  Participants
    number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 16
    Female | 2 | 0 | 1 | 0 | 0 | 3
    Male | 1 | 4 | 2 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Stage I - Safety (Type, Frequency, Severity and Relationship of Adverse Events to Study Treatment) and Tolerability
Description: Determine the maximum tolerated dose (MTD) of lenalidomide when given in combination with rituximab, Ifosfamide, etoposide, and carboplatin (RICE) for the treatment of DLBCL patients in first relapse by incidence of dose-limiting toxicity (DLT) for Stage I Patients Only
Time Frame: Cycle 1 of Treatment (28 Days)
Measure: Number; unit: mg
Groups:
- Revlimid (Lenalidomide) in Combination: Study of Lenalidomide in Combination with Rituximab, Ifosphamide, Etoposide, and Carboplatin (RICE-R) as Salvage Therapy with Single Agent Lenalidomide as Maintenance Therapy Post-Autologous Stem Cell Transplantation
  Revlimid: Stage I:
  Cohort 1: RICE + Lenalidomide 10mg days 1-7 Cohort 2: RICE + Lenalidomide 15mg days 1-7 Cohort 3: RICE + Lenalidomide 20mg days 1-7 Cohort 4: RICE + Lenalidomide 25mg days 1-7
  Stage II:
  RICE + Lenalidomide at the MTD days 1-7
  Stage III:
  Lenalidomide 25mg days 1-21 every 28 days
Arm/Group | Revlimid (Lenalidomide) in Combination
Number analyzed (Participants) | 13
mg | 25

2. Primary Outcome: Stage II - Overall Response Rate
Description: Rate of overall response by incidence of Complete Response, Partial Response, and Stable Disease per Modified International Working Group (IWG) response criteria for patients enrolled in Stage II
Time Frame: After 2 Cycles of Treatment (28 Day Cycles)
Population: Only patients enrolled in Stage II analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
Participants | 0 | 0 | 0 | 0 | 2

3. Primary Outcome: Stage III - Overall Response Rate
Description: Rate of overall response by incidence of Complete Response, Partial Response, and Stable Disease per Modified International Working Group (IWG) response criteria for patients enrolled in Stage III
Time Frame: After 2 Cycles of Treatment (28 Day Cycles)
Population: No Stage III Participants Enrolled
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Stage I - Dose Limiting Toxicity Incidence Rate
Description: Incidence of DLT in patients enrolled in stage I for determination of MTD
Time Frame: Cycle 1 of Treatment (28 Days)
Population: Rate of DLTs occurred in Stage I Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 0
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Stage II - 1 Year Progression Free Survival (PFS)
Description: Rate of Progression Free Survival (PFS) at 1 Year of patients enrolled in stage II
Time Frame: Up to 1 Year
Population: Only patients enrolled in Stage II analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
Participants | 0 | 0 | 0 | 0 | 2

6. Secondary Outcome: Stage II - 2 Year Progression Free Survival (PFS)
Description: Rate of Progression Free Survival (PFS) at 1 Year of patients enrolled in stage II
Time Frame: Up to 2 Years
Population: Only patients enrolled in Stage II analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
Participants | 0 | 0 | 0 | 0 | 2

7. Secondary Outcome: Stage II - 1 Year Overall Survival (OS)
Description: 1 Year Overall Survival (OS) of patients enrolled in stage II
Time Frame: Up to 1 Year
Population: Only patients enrolled in stage II analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
Participants | 0 | 0 | 0 | 0 | 2

8. Secondary Outcome: Stage II - 2 Year Overall Survival (OS)
Description: 2 Year Overall Survival (OS) of patients enrolled in stage II
Time Frame: Up to 2 years
Population: Only patients enrolled in stage II analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
Participants | 0 | 0 | 0 | 0 | 2

9. Secondary Outcome: Stage III - Progression Free Survival (PFS) Rate Post Transplant
Description: Rate of Progression Free Survival (PFS) 2 years post Transplant
Time Frame: 2 Years Post Transplant
Population: No Stage III Participants Enrolled
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Stage III - Overall Survival (OS)
Description: 2 Year Overall Survival (OS) of patients enrolled in stage III
Time Frame: 2 Years Post Transplant
Population: No Stage III Participants Enrolled
Arm/Group | Stage I, Cohort 1 | Stage I, Cohort 2 | Stage I, Cohort 3 | Stage I, Cohort 4 | Stage II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Adverse Events were collected irrespective of dose level and therefore cannot be reported by dose level
Groups:
- RICE + Lenalidomide: RICE + Lenalidomide days 1-7
Arm/Group | RICE + Lenalidomide
All-Cause Mortality (participants affected / at risk) | 2/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RICE + Lenalidomide (N=16)
RSV Infection (Infections and infestations) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1)
Secondary Primary Malignancy (+MDS) (Blood and lymphatic system disorders) | 1 (1)
Infectious Enterocolitis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fever (absence of neutropenia) (Investigations) | 2 (2)
Sepsis (Gram Positive) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RICE + Lenalidomide (N=16)
Neuropathy (Nervous system disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 2
Anemia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 10

LIMITATIONS AND CAVEATS:
Adverse Events were collected irrespective of dose level and therefore cannot be reported by dose level. A portion of the Stage II patients were enrolled at an external site and some demographic details of these patients are no longer available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes